CLINICAL TRIAL: NCT00589771
Title: Clinical and Cytokine Response to Saccharomyces Boulardii Therapy in Diarrhea Dominant Irritable Bowel Syndrome
Brief Title: Saccharomyces Boulardii in Irritable Bowel Syndrome
Acronym: SB-IBS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Biocodex (Industry)
Responsible Party: Principal Investigator, Zaigham Abbas, Consultant Gastroenterologist, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 674- MED; 2007-674MED-ERC; SB-IBS-674; SB-IBS-cytokines-674
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Diarrhea Dominant Irritable Bowel Syndrome
Keywords: IBS; Saccharomyces boulardii; probiotics; cytokine; histology; Efficacy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): 1. Capsule Saccharomyces boulardii 250 mg TDS for six weeks.
  2. Ispahgula husk 1 Tsf daily after dinner for six weeks.
  Interventions: Drug: Saccharomyces boulardii
- B (Placebo Comparator): 1. Capsule Placebo TDS for six weeks.
  2. Ispaghula husk 1 Tsf daily after dinner for six weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saccharomyces boulardii — 1. Saccharomyces boulardii one capsule 250mg TDS for 6 weeks
  2. Ispaghula husk 1 Tsf daily after dinner for six weeks
  Other Names: Enflor
  Arms: A
Drug: Placebo — 1. Cap Placebo TDS for six weeks
  2. Ispaghula husk 1 Tsf daily after dinner for six weeks
  Arms: B

SUMMARY:
Various studies have been conducted in past using different strains of probiotics in evaluating IBS symptoms. The results are by no means consistent and the overall impact of probiotics in IBS remains unclear. However, recently O'Mahony L et al have shown that Bifidobacterium infantis 35624 alleviates symptoms in IBS; this symptomatic response was associated with normalization of the ratio of an anti-inflammatory to a proinflammatory cytokine (IL-10/IL-12 ratio), suggesting an immune-modulating role for this organism, in this disorder.Saccharomyces boulardii is a probiotic yeast that has been successfully used for the antibiotic induced diarrhea, prevent relapse of Clostridium difficile and Crohn's disease. It ameliorates intestinal injury and inflammation caused by a wide variety of enteric pathogens.We therefore plan a Double-blind, randomized, placebo-controlled study to assess the effects of Saccharomyces boulardii in improving symptomatology of diarrhea predominant IBS and its effect on quality of life. We also plan to assess the changes in the relative production of anti-inflammatory interleukin (IL)-10 to proinflammatory cytokines (IL-12, IL-8 and TNFα).

ELIGIBILITY:
Inclusion Criteria:

1. Diarrhea-predominant IBS satisfying ROME III criteria.
2. Adults aged 18-70

Exclusion Criteria:

1. Pregnant and lactating females
2. Inflammatory bowel disease and other systemic disease
3. Patients on anti-diarrheal and antibiotics drugs
4. Patients with any ongoing infection
5. Not willing to participate
6. Allergy to any of Saccharomyces boulardii components
7. Central venous catheter carriers
8. Other probiotics e.g., Lactobacillus and Bifidobacterium

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of Saccharomyces boulardii in reducing clinical symptoms, improving cytokines levels and histology features | 6 weeks

SECONDARY OUTCOMES:
Assess the efficacy of Saccharomyces boulardii in improving quality of life and safety of the drug | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zaigham Abbas, FACG, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan